CLINICAL TRIAL: NCT06510608
Title: Evaluation of the Roles of Salivary Mitofusin-1 and Mitofusin-2 Levels in Periodontal Disease
Brief Title: Periodontal Disease and Salivary Mitofusin Levels
Status: Not yet recruiting | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Okumuş, Assistant Professor, Erzincan University
Other Study IDs: EUDF-OKUMUS-004
Record Dates: First submitted 2024-07-05; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis; Periodontal Diseases; Gingivitis
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — human saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy
  Interventions: Diagnostic Test: Biochemical analysis of saliva sample
- Gingivitis
  Interventions: Diagnostic Test: Biochemical analysis of saliva sample
- Periodontitis
  Interventions: Diagnostic Test: Biochemical analysis of saliva sample

INTERVENTIONS:
Diagnostic Test: Biochemical analysis of saliva sample — It is the examination of saliva samples taken with biochemical methods. In this way, the substances in its content and the concentration of cytokines are analyzed.

SUMMARY:
The aim of this observational study is to find out whether there is a level difference in salivary mitofusin-1 and mitofusin-2 levels due to changes in periodontal status. The main question it aims to answer is:

* Do salivary mitofusin-1 and mitofusin-2 levels of periodontitis patients differ from healthy patients?
* Could salivary mitofusin-1 and mitofusin-2 levels be biomarkers for periodontal disease?

Biochemical analysis will be performed on saliva samples taken at once from gingivitis or periodontitis patients and healthy individuals who apply to the periodontology clinic, at the initial stage of the treatment. There is no ongoing monitoring or second sampling.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65.
* Willing to participate in the study and provide a saliva sample.
* Having a healthy periodontal condition, gingivitis, or periodontitis (Stage 3-4, Grade C).
* Having fasted from any food or drink (except water) for the past 2 hours prior to providing the saliva sample.
* Having refrained from brushing teeth or using mouthwash in the past 2 hours prior to providing the saliva sample.
* Not having any systemic diseases.
* Not currently taking any medications regularly.

Exclusion Criteria:

* Having used antibiotics within the last 6 months.
* Having received periodontal treatment within the last 6 months.
* Having fewer than 20 teeth (excluding third molars).
* Having any systemic diseases.
* Not smoking or having quit at least 5 years ago.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gingivitis and periodontitis presenting to the periodontology clinic, as well as healthy individuals
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Mitofusin-1 concentration | Up to four weeks from start of work
  Mitofusin-1 concentration in saliva, determined as a result of biochemical analysis
Mitofusin-2 concentration | Up to four weeks from start of work
  Mitofusin-2 concentration in saliva, determined as a result of biochemical analysis
IL-1B concentration | Up to four weeks from start of work
  IL-1B concentration in saliva, determined as a result of biochemical analysis

REFERENCES:
- [Derived] Okumus OF, Kurt N, Kantarci A. Salivary mitofusin levels in periodontal disease: a cross-sectional case-control study. BMC Oral Health. 2025 Oct 6;25(1):1542. doi: 10.1186/s12903-025-06932-0. PMID 41053720